CLINICAL TRIAL: NCT00280384
Title: An Electrophysiological Study Of E2014 In Healthy Adult Male Japanese And Caucasian Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Limited (Industry)
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E2014-J081-133
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Results first posted 2013-04-25 (Estimated); Last update posted 2013-04-25 (Estimated); Status verified 2013-04

CONDITIONS: Spasmodic Torticollis
MeSH Terms: conditions — Torticollis | interventions — rimabotulinumtoxinB

ARMS (2):
- E2014 (Botulinum toxin type B) (Active Comparator)
  Interventions: Drug: E2014 (Botulinum toxin type B)
- E2014 (Botulinum toxin type B) Placebo (Placebo Comparator)
  Interventions: Drug: E2014 (Botulinum toxin type B) Placebo

INTERVENTIONS:
Drug: E2014 (Botulinum toxin type B) — A single-dose injection solution containing 20 units (U), 100 U, or 500 U/ 0.2 milliliters (mL) of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese and Caucasian participants. Duration of treatment lasted for 12 weeks: from Day -1 to Week 12. Participants were hospitalized from a day before study treatment to Day 8 for 9 nights and 10 days, and visited at the medical institution on Days 10 and 14, and Weeks 4 and 12.
  Arms: E2014 (Botulinum toxin type B)
Drug: E2014 (Botulinum toxin type B) Placebo — A single-dose injection solution of E2014 Placebo was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese and Caucasian participants. Duration of treatment lasted for 12 weeks: from Day -1 to Week 12. Participants were hospitalized from a day before study treatment to Day 8 for 9 nights and 10 days, and visited at the medical institution on Days 10 and 14, and Weeks 4 and 12.
  Arms: E2014 (Botulinum toxin type B) Placebo

SUMMARY:
To evaluate inter-ethnic similarity in pharmacodynamics between Japanese and Caucasian healthy adult male subjects by comparing electrophysiological reactions after administering E2014 to extensor digitorum brevis muscle (EDB).

ELIGIBILITY:
Inclusion criteria:

1. Participants aged between 20 and 44 years at the time of obtaining informed consent.
2. Participants whose M wave amplitude potential (between baseline and negative peak) in the EDB by stimulating peroneal nerve in the foot joints is 1 mV or more during electrophysiological examinations at the times of screening and immediately before administration.
3. Participants who are judged to be eligible for study entry by an investigator or subinvestigator at screening and at immediately before pre-treatment medical examination.
4. Participants who are given a full explanation about the objective and details of this study before starting screening and give written consent based on their free will.

Exclusion Criteria:

1. Participants who have a complication or history of peripheral neuropathy, nerve root impairment, muscle disease.
2. Participants with a disease that may influence the study drug evaluation, such as disorders of the gastrointestinal tract, liver, respiratory, endocrine, hematological, neurological, psychiatric and cardiovascular system, and congenital abnormality in metabolism.
3. Participants who have accessory deep peroneal nerve.
4. Participants who previously received a treatment with botulinum toxin.
5. Participants with a history of hypersensitivity to any component of E2014 (human serum albumin, succinate buffer solution).
6. Participants who are positive for urine drug screening at the time of screening or immediately before study drug administration.
7. Participants who received prescription drug(s) within 1 month before study drug administration.
8. Participants who have been treated with another investigational drug within 4 months before study drug administration.
9. Participants who have experienced heavy exercise or hard labor within 2 weeks before study drug administration.
10. Participants who underwent blood transfusion within 3 months before, those whose 400 mL of whole blood was collected within 3 months before, or those whose 200 mL of whole blood was collected within 1 month before study drug administration.
11. Participants who are positive for hepatitis B surface antigen (HBs antigen), hepatitis C virus (HCV) antibody, or serologic test for syphilis (STS).
12. Participants who received a diagnosis of acquired immunodeficiency syndrome (AIDS) or those with positive result for human immunodeficiency virus.
13. Participants who are unwilling or unable to abide by the requirements of this study, or those who may violate the prohibitions and restrictions of this study.
14. Participants who are judge to be ineligible for study entry by a principal investigator or subinvestigator.

Ages: 20 Years to 44 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hiroki Shimizu, Study Director — Eisai Co., Ltd.
Locations (1):
- Kagoshima, Kagoshima-ken, Japan

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 94 participants screened (60 Japanese, 34 Caucasian), 57 (29 Japanese and 28 Caucasian) participants were admitted to the hospital. 9 (5 Japanese and 4 Caucasian) participants did not receive the study drug. 48 participants received the study drug (24 Japanese and 24 Caucasian) and were considered the treated population.
Groups:
- E2014 (Botulinum Toxin Type B) Placebo- Japanese: A single-dose injection solution of E2014 Placebo was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese participants.
- E2014 (Botulinum Toxin Type B) 20 U - Japanese: A single-dose injection solution containing 20 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese participants.
- E2014 (Botulinum Toxin Type B) 100 U - Japanese: A single-dose injection solution containing 100 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese participants.
- E2014 (Botulinum Toxin Type B) 500 U - Japanese: A single-dose injection solution containing 500 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Japanese participants.
- E2014 (Botulinum Toxin Type B) Placebo - Caucasian: A single-dose injection solution of E2014 Placebo was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Caucasian participants.
- E2014 (Botulinum Toxin Type B) 20 U - Caucasian: A single-dose injection solution containing 20 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Caucasian participants.
- E2014 (Botulinum Toxin Type B) 100 U - Caucasian: A single-dose injection solution containing 100 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Caucasian participants.
- E2014 (Botulinum Toxin Type B) 500 U - Caucasian: A single-dose injection solution containing 500 U/ 0.2 mL of E2014 was administered to extensor digitorum brevis (EDB) muscle in the left lower limb to Caucasian participants.
Period: Overall Study
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Started | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48
Age Continuous [Mean (Standard Deviation); unit: years] | 22.7 (2.9) | 28.0 (5.4) | 23.3 (2.9) | 22.2 (2.6) | 33.7 (2.7) | 34.5 (3.7) | 32.7 (2.9) | 29.3 (2.6) | 28.3 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 48

OUTCOME MEASURES:

1. Primary Outcome: Maximum Rates of Extensor Digitorum Brevis (EDB) Muscle M-Wave Amplitude Reduction From Baseline
Description: The pharmacodynamic effect of botulinum toxin type B (E2014) was evaluated based on the inhibition of EDB M-wave amplitude induced by stimulation of the deep peroneal nerve in the left ankles of the study participants. EDB M-wave amplitudes (mV) were measured at screening (baseline), and Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, Day 14, Week 4, and Week 12. Rates of EDB M-wave amplitude reduction from baseline were then calculated at each time point. The maximum rates of EDB M-wave amplitude reduction from baseline were presented as a percentage.
Time Frame: Baseline and Up to Week 12
Measure: Mean (Standard Deviation); unit: Percentage of Reduction
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of Reduction | 9.02 (13.51) | 48.53 (16.98) | 70.95 (6.12) | 81.62 (7.55) | 14.33 (9.05) | 42.77 (20.78) | 50.70 (9.35) | 74.47 (6.56)

2. Primary Outcome: Extensor Digitorum Brevis (EDB) Muscle M-Wave Amplitude at Baseline
Description: The pharmacodynamic effect of botulinum toxin type B (E2014) was evaluated based on the inhibition of EDB M-wave amplitude induced by stimulation of the deep peroneal nerve in the left ankles of the study participants. EDB M-wave amplitudes (mV) were measured at screening (baseline).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: EDB M-Wave Amplitude at Baseline (mV)
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
EDB M-Wave Amplitude at Baseline (mV) | 6.67 (1.25) | 4.73 (1.13) | 4.95 (1.48) | 4.78 (1.70) | 7.12 (1.40) | 5.48 (1.92) | 6.00 (2.52) | 5.12 (1.15)

3. Primary Outcome: Maximum Rates of Extensor Digitorum Brevis (EDB) Muscle M-Wave Area Reduction From Baseline
Description: The pharmacodynamic effect of botulinum toxin type B (E2014) was evaluated based on the inhibition of EDB M-wave area induced by stimulation of the deep peroneal nerve in the left ankles of the study participants. EDB M-wave area (mVms) was measured at screening (baseline), and Day 1, Day 2, Day 4, Day 6, Day 8, Day 10, Day 14, Week 4, and Week 12. Rates of EDB M-wave area reduction from baseline were then calculated at each time point. The maximum rates of EDB M-wave area reduction from baseline were presented as a percentage.
Time Frame: Baseline and Up to 12 Weeks
Measure: Mean (Standard Deviation); unit: Percentage of Reduction
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
Percentage of Reduction | 13.13 (17.19) | 43.22 (15.50) | 74.97 (7.60) | 79.03 (8.85) | 14.98 (12.06) | 45.65 (20.34) | 48.12 (11.09) | 75.65 (4.72)

4. Primary Outcome: Extensor Digitorum Brevis (EDB) Muscle M-Wave Area At Baseline
Description: The pharmacodynamic effect of botulinum toxin type B (E2014) was evaluated based on the inhibition of EDB M-wave area induced by stimulation of the deep peroneal nerve in the left ankles of the study participants. EDB M-wave area (mVms) was measured at screening (baseline).
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: EDB M-Wave Area at Baseline (mVms)
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 6 | 6 | 6
EDB M-Wave Area at Baseline (mVms) | 18.90 (4.23) | 14.97 (3.80) | 14.38 (4.67) | 14.85 (4.78) | 18.68 (1.99) | 16.18 (4.03) | 17.57 (5.67) | 14.58 (2.09)

ADVERSE EVENTS:
Arm/Group | E2014 (Botulinum Toxin Type B) Placebo- Japanese | E2014 (Botulinum Toxin Type B) 20 U - Japanese | E2014 (Botulinum Toxin Type B) 100 U - Japanese | E2014 (Botulinum Toxin Type B) 500 U - Japanese | E2014 (Botulinum Toxin Type B) Placebo - Caucasian | E2014 (Botulinum Toxin Type B) 20 U - Caucasian | E2014 (Botulinum Toxin Type B) 100 U - Caucasian | E2014 (Botulinum Toxin Type B) 500 U - Caucasian
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 1/6 | 0/6 | 0/6 | 1/6 | 0/6 | 0/6 | 2/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | E2014 (Botulinum Toxin Type B) Placebo- Japanese (N=6) | E2014 (Botulinum Toxin Type B) 20 U - Japanese (N=6) | E2014 (Botulinum Toxin Type B) 100 U - Japanese (N=6) | E2014 (Botulinum Toxin Type B) 500 U - Japanese (N=6) | E2014 (Botulinum Toxin Type B) Placebo - Caucasian (N=6) | E2014 (Botulinum Toxin Type B) 20 U - Caucasian (N=6) | E2014 (Botulinum Toxin Type B) 100 U - Caucasian (N=6) | E2014 (Botulinum Toxin Type B) 500 U - Caucasian (N=6)
White Blood Cell Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Aspartate Aminotransferase Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Eosinophil Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neutrophil Increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Neck Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No